CLINICAL TRIAL: NCT07055542
Title: Creating A RIsk Assessment Biomarker Tool to Prevent Seasonal and Thunderstorm Asthma: The CARISTA Study
Brief Title: Creating A Risk Assessment Tool for Thunderstorm Asthma: the CARISTA Study
Acronym: CARISTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: The Alfred (Other); Eastern Health (Other); Austin Hospital, Melbourne Australia (Other); Monash Medical Centre (Other); Queensland University of Technology (Other); Northern Hospital, Australia (Other); Western Hospital, Australia (Other Government); Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CT31402
Record Dates: First submitted 2025-06-10; First posted 2025-07-09 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-06

CONDITIONS: Allergic Asthma; Thunderstorm Asthma; Seasonal Allergic Rhinitis; Grass Pollen Allergy; Asthma Exacerbation Due to Thunderstorm; Asthma Acute
Keywords: asthma; allergy; grass pollen allergy; ryegrass pollen; prospective symptom monitoring; seasonal allergic rhinitis; hay fever; seasonal allergic rhinoconjunctivitis; serum specific IgE; spirometry
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Asthma; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Prospective cohort study to undertake risk prediction modelling for seasonal allergic and thunderstorm asthma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observational (Other): prospective observational cohort
  Interventions: Diagnostic Test: Observational

INTERVENTIONS:
Diagnostic Test: Observational — Prospective observational study

SUMMARY:
Thunderstorm asthma is a recurring public health emergency in South-Eastern Australia which occurs in springtime. The major identified risk factors for thunderstorm asthma is hay fever and allergy to ryegrass pollen. The goal of the CARISTA study is to identify the risk of springtime allergic and thunderstorm asthma in allergic adults living in South-Eastern Australia. To do this the investigators will recruit 530 people who have hay fever and test them for allergy to ryegrass pollen and undertake simple lung function testing. The investigators will ask study participants to complete a customised symptom tracker over the springtime pollen season for 2 consecutive years. The outcome the investigators are looking for is an asthma exacerbation or worsening asthma symptoms. This study will enable the investigators to identify indicators (biomarkers) of severe and moderate asthma exacerbations in order to identify those at risk of thunderstorm and seasonal asthma so protective treatments and strategies can be advised.

DETAILED DESCRIPTION:
Thunderstorm asthma is a recurring public health emergency in South-Eastern Australia with increasing risks due to climate change. Yet thunderstorm asthma is only the "tip of the iceberg" of documented seasonal surges in emergency asthma presentations due to ryegrass pollen allergy - an escalating challenge to healthcare provision in South-Eastern Australia. The CARISTA (Creating A Risk assessment biomarker tool to prevent Seasonal allergic and Thunderstorm Asthma) study aims to address these profound health impacts.

The CARISTA study will recruit adults at high risk of seasonal allergic asthma and thunderstorm asthma who will be monitored using a customised secure data platform for asthma and allergic rhinitis symptoms over two consecutive spring seasons (2025/2026/2027). Participants with self-reported or diagnosed seasonal allergic rhinitis and/or seasonal allergic asthma will be recruited before springtime and their baseline allergic rhinitis and/or asthma symptoms, respiratory function and blood biomarkers (allergy or sensitisation to ryegrass pollen, levels of inflammatory cells [eosinophils]) will be measured.

The key symptoms of interest are moderate or severe asthma exacerbations which are defined as an increase in asthma symptoms requiring intervention with an emergency medical visit, use of oral corticosteroid therapy or of regular preventive asthma therapy. These asthma exacerbations will be used to establish a biomarker-based estimate of risk for seasonal allergic asthma exacerbations to inform preventive clinical practice. The key biomarker will be the threshold of serum specific IgE (sp-IgE) to ryegrass pollen and its allergen sub-components, but other biomarkers such as lung function, eosinophil levels, and allergen component sensitisation will be simultaneously assessed.

This study brings together a team of world-leading multidisciplinary and cross-sectoral clinicians and researchers in Respiratory Medicine, Allergy, Primary Health Care, Epidemiology, Public Health, Statistical modelling and Botany from multiple health and academic institutions.

Overall, CARISTA will test a new approach to predict risk for seasonal allergic asthma to identify treatable traits for preventing seasonal allergic asthma exacerbations to reduce the recurrent annual health threat of seasonal and thunderstorm asthma, address community and health care provider concerns and uncertainty regarding preventive treatment and management.

ELIGIBILITY:
Inclusion Criteria:

Consenting adults aged 18 to 70 years with seasonal allergic rhinitis

willing to undertake:

* Lung function testing
* Blood sample collection for risk factor identification, -Prospectively logging their symptoms and medications through the springtime season using the CARISTA symptom monitoring platform . -

Exclusion Criteria:

* Individuals unable to provide informed consent
* Individuals who do not suffer from symptoms of seasonal allergic rhinitis
* Individuals who do not consent to lung function testing and blood sample collection - Individuals with unstable asthma (FEV1 by spirometry less than 70% predicted), a recent exacerbation or change of asthma preventive medication use (within one month) would be excluded, although re-screening would be permitted after one month, time permitting.
* Individuals with severe asthma requiring the use of continuous oral corticosteroids or biological medication for severe asthma.
* The presence of any medical illness, such as cardiac disease, pre-existing illness or immunomodulatory therapy that, in the opinion of the Investigators, would compromise participant safety or the derivation of biomarkers during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation of gender identify
Enrollment: 530 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Moderate or Severe Asthma Exacerbations | Over 13 weeks from 1 October - 31 December
  Moderate and/or severe asthma exacerbations determined by
  * increased rescue bronchodilator medication use to a minimum of 4 puffs/day and doubling of baseline use, for 2 consecutive days
  * an increase in asthma symptoms requiring institution of, or doubling the regular dose of preventer asthma therapy
  * asthma symptoms requiring oral corticosteroid therapy
  * institution of emergency asthma treatment or medical attendance for emergency asthma treatment indicative of uncontrolled asthma.

SECONDARY OUTCOMES:
Number of Participants with Severe asthma exacerbations | Over 13 weeks from 1 October - 31 December
  Institution of emergency asthma treatment or medical attendance for emergency asthma treatment indicative of uncontrolled asthma or institution of oral corticosteroid therapy for asthma by a medical practitioner.
Number of Participants with Onset of uncontrolled asthma | Over 13 weeks from 1 October - 31 December
  Onset of uncontrolled asthma determined by a worsening of asthma symptoms measured by the Asthma Control Questionnaire (ACQ-5:) increasing by 0.5 from baseline and being greater than 1.5. The minimum value = 0 and maximum value = 30. Higher scores indicate worse asthma symptoms.

OTHER OUTCOMES:
Number of Participants with Rhinitis symptoms | Over 13 weeks from 1 October - 31 December
  Recorded on Total Nasal Symptom Score (TNSS). The minimum value = 0 and maximum value = 9. Higher scores indicate more and worse rhinitis symptoms.
Number of Participants with Hospital presentations for asthma | Over 13 weeks from 1 October - 31 December
  Hospital emergency attendance for worsening of acute asthma
Number of Participants with Emergency attendance for asthma care | Over 13 weeks from 1 October - 31 December
  Emergency attendance to a clinical facility for acute asthma care

CONTACTS AND LOCATIONS:
Overall Officials: Jo A Douglass, MD, Study Chair — University of Melbourne & Royal Melbourne Hospital; Phillip Bardin, MD, Principal Investigator — Hudson Institute of Medical Research; Frank Thien, MD PhD, Principal Investigator — Eastern Health; Mark Hew, MD PhD, Principal Investigator — The Alfred
Locations (1):
- The Royal Melbourne Hospital, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT07055542/Prot_SAP_000.pdf
  • Informed Consent Form: Informed Consent (2025-01-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT07055542/ICF_001.pdf